CLINICAL TRIAL: NCT04976712
Title: Core Temperature in Patients With Out of Hospital Cardiac Arrest in South Tyrol - a Prospective Observational Study
Brief Title: Core Temperature in Patients With OHCA
Acronym: CT-OCHA
Status: Recruiting | Type: Observational
Sponsor: Azienda Sanitaria dell'Alto Adige (Other)
Collaborators: Institute of Mountain Emergency Medicine (Other)
Responsible Party: Principal Investigator, Elisabeth Gruber, Principal Investigator, Azienda Sanitaria dell'Alto Adige
Other Study IDs: BZ-107-2020
Record Dates: First submitted 2021-06-23; First posted 2021-07-26 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Out-Of-Hospital Cardiac Arrest; Accidental Hypothermia; Temperature Change, Body
Keywords: Out-Of-Hospital Cardiac Arrest; Accidental Hypothermia; Core Temperature
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Hypothermia; Body Temperature Changes

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A prospective observational study aiming to monitor core temperature via an esophageal probe in out of hospital cardiac arrest during transport and until arrival in hospital. Insertion of an esophageal temperature probe will be done on scene during ongoing resuscitation manoeuvres based on European Resuscitation Council Guidelines 2015 (or newer). Environmental temperature influence and hypothermia prevention interventions will be monitored.

DETAILED DESCRIPTION:
Prospective observational study to evaluate the body temperature difference in patients in out of hospital cardiac arrest on site and at arrival at the hospital.

If the patient fulfills the inclusion criteria and after establishment of CPR measures according the ERC resuscitation guidelines (2015 or newer) an esophageal probe will be inserted and bodytemperature is measured; on site ambiental temperature will also be measured. Weather conditions, altitude on site, activity of the patient and hypothermia protection (eg. clothes) will bei documented. On arrival in hospital the body temperature will be measured with the esophageal probe;

ELIGIBILITY:
Inclusion Criteria:

* Out of hospital cardiac arrest
* Patients transferred to hospital
* > 18 years

Exclusion Criteria:

* Obvious signs of death
* Obvious lethal injury/injuries incompatible with life
* Confirmation of death on scene
* < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with out of hospital cardiac arrest transferred to hospital
Sampling Method: Probability Sample
Enrollment: 256 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Core temperature at hospital arrival | through study completion, an average of 1 year
  ° Celsius

SECONDARY OUTCOMES:
Core temperature at ROSC | through study completion, an average of 1 year
  ° Celsius
Environmental temperature on scene | through study completion, an average of 1 year
  ° Celsius
Time of resuscitation from OHCA to ROSC | through study completion, an average of 1 year
  minutes
OHCA rhythm at arrival of ALS team | through study completion, an average of 1 year
  ECG rhythm: asystolia, PEA, ventricular fibrillation, ventricular tachicardia
Use of mechanical chest compression device on prehospital intervention | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rosmarie Oberhammer, MD, Study Director — Azienda Sanitaria dell'Alto Adige
Locations (1):
- Bruneck Regional Hospital, Bruneck, Italy